CLINICAL TRIAL: NCT04948099
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of VIB1116 in Conventional Dendritic Cell (cDC) and Plasmacytoid Dendritic Cell (pDC)-Mediated Rheumatic Diseases
Brief Title: A Study of Single and Multiple Ascending Doses of VIB1116 in Rheumatic Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIB1116.P1.S1
Record Dates: First submitted 2021-06-16; First posted 2021-07-01 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Dendritic Cell -Mediated Rheumatic Diseases
Keywords: Autoimmune disease; Rheumatic disease; Phase 1
MeSH Terms: conditions — Autoimmune Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIB1116 (Experimental): Single dose of VIB1116, SC or IV administration.
  Multiple doses of VIB1116, SC administration.
  Interventions: Drug: VIB1116
- Placebo (Placebo Comparator): Single dose of Placebo, SC or IV administration.
  Multiple doses of Placebo, SC administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIB1116 — VIB1116
  Arms: VIB1116
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A first-in-human study to evaluate the safety and tolerability of escalating, single and multiple ascending doses of VIB1116 in adult participants with rheumatic diseases.

DETAILED DESCRIPTION:
Study acquired from Horizon in 2024. Originally Viela Bio was the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age and ≤ 60 years of age and a body mass index (BMI) < 30 kg/m² or, in patients who have completed dosing with a vaccine against COVID-19 and are at least 1 month post the last dose, ≤ 65 years of age and BMI < 35 kg/m^2
* A diagnosis of one of a specified list of rheumatologic diseases at least 6 months prior to screening.
* Stable dosing (or no use) of glucocorticoid or disease-modifying antirheumatic drugs (DMARDs) used for treatment of rheumatologic disease for ≥ 28 days prior to randomization.
* Willing to practice study-required contraception.

Exclusion Criteria:

* Planning to change treatment for rheumatologic disorder within 4 months after randomization
* Known immunodeficiency disorder or history of splenectomy, organ or cell-based transplantation, total lymphoid irradiation or T-cell vaccination or transfusion in prior 6 months
* Treatment with prednisone or equivalent at a dose > 10 mg/day or intraarticular, intravenous or intramuscular steroids within 28 days prior to screening
* Treatment with any of the following medications within 28 days prior to screening (unless otherwise specified below) above the given doses:

  * Mycophenolate mofetil > 2 g/day
  * Methotrexate > 20 mg/week
  * Leflunomide > 20 mg/day within 6 months prior to screening or receipt of leflunomide in combination with any dose of methotrexate
  * Azathioprine > 2 mg/kg/day
  * Cyclosporine (except eye drops); tacrolimus (except topical), sirolimus, thalidomide, lenalidomide, 6-mercaptopurine, or voclosporin
  * Hydroxychloroquine > 400 mg/day
  * Chloroquine > 250 mg/day
  * Quinacrine > 100 mg/day
  * Sulfasalazine > 3 g/day, except that no more than 1 g/day is permitted if used in combination with methotrexate
  * Dapsone > 100 mg/day
  * Danazol > 800 mg/day
  * Any other nonbiologic immunosuppressive/immunomodulatory agent not already specified (eg, mizoribine, retinoids, adrenocorticotropic hormone analogs, dehydroepiandrosterone [DHEA]) within 2 weeks prior to screening.
  * Receipt of any biologic B cell-depleting therapy within 12 months or non-depleting B cell-directed therapy within 6 months
  * Receipt of abatacept, etanercept, or other biologic immunomodulatory agent or immunoglobulins within 3 months
  * Receipt of any other biologic disease modifying antirheumatic drug (bDMARD) not already specified, such as any targeted therapy (other than Janus kinase [JAK] inhibitor), or receipt of cyclophosphamide or chlorambucil within 6 months
  * Receipt of JAK inhibitors within 3 months
  * Receipt of anticoagulants other than anti-platelet drugs in prior 28 days
  * Active malignancy, history of malignancy within prior 10 years (limited exceptions) or known first degree relative with a hereditary cancer syndrome unless the patient is known to be free of the predisposing genetic mutation
  * Receipt of live vaccine or live therapeutic infectious agent within the 28 days prior to screening.
  * Pregnancy, lactation, or planning to become pregnant or donate/retrieve eggs before the end of study follow-up.
* Hepatitis B or C infection, HIV infection, evidence of active TB or being at high risk for TB
* History of any severe herpes virus infection (including any history of severe Epstein-Barr virus, cytomegalovirus disease, end-organ disease, disseminated herpes simplex, disseminated zoster, or ophthalmic zoster) or > 1 episode of herpes zoster in the 2 years prior to screening and/or any opportunistic infection in the prior 2 years
* Infection requiring parenteral antimicrobial therapy within 60 days of screening or any clinically significant active or suspected infection ( within 28 days prior to screening
* History of anaphylaxis to any human immunoglobulin therapy or monoclonal antibody.
* Blood tests at screening (performed in the central laboratory) that meet study requirements including but not limited to normal coagulation testing and glomerular filtration rate < 50 mL/min/1.73
* High risk for COVID-19 or for severe COVID-19

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events, treatment-emergent serious adverse events, and adverse events of special interest | Up to Day 141

SECONDARY OUTCOMES:
Serum concentration of VIB1116 and noncompartmental PK parameters | Up to Day 141
Change from baseline in the blood levels of plasmacytoid dendritic cells | Up to Day 141
Percentage of Participants who are ADA (antidrug antibody) positive | Up to Day 141
Titer in ADA positive participants | Up to Day 141

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (8):
  - Pinnacle Research Group, Anniston, Alabama
  - Clinical Research of W FL, Clearwater, Florida
  - Jacksonville Clinical Research, Jacksonville, Florida
  - Accurate Clinical Research, Lake Charles, Louisiana
  - Altoona Clinical Research, Duncansville, Pennsylvania
  - Rheumatology Associates, Dallas, Texas
  - SW Rheumatology Center, Mesquite, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
- Poland (3):
  - Klinika Reumatologii i Rehabilitacji Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im W. Degi, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - ARS RHEUMATICA Sp. z o.o. REUMATIKA-Centrum Reumatologii NZOZ, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: No